CLINICAL TRIAL: NCT03595800
Title: Extension of a Phase III Randomized Study of Allogeneic Hematopoietic Stem Cell Transplantation From One Haplotype Mismatch Related Donor or From an Unrelated Donor to Younger Patients Eligible for Reduced-intensity Conditioning Regimen-HaploMUD-RIC-01
Brief Title: Extension of a Study of Allogeneic Hematopoietic Stem Cell Transplantation From One Haplotype Mismatch Related Donor or From an Unrelated Donor to Younger Patients Eligible for Reduced-intensity Conditioning Regimen
Acronym: HaploMUD-RIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaploMUD-RIC-01
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2021-03

CONDITIONS: Acute Leukemia; Non Hodgkin Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- haploidentical related donors (Experimental)
  Interventions: Procedure: Hematopoietic stem cells transplantation
- Matched unrelated donor (Active Comparator)
  Interventions: Procedure: Hematopoietic stem cells transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cells transplantation — Allogeneic Hematopoietic stem cells transplantation

SUMMARY:
This study is an extension to younger patients of the currently ongoing national, multicenter, open-label, randomized phase III HAPLOMUDELDERLY which evaluates elderly patients with hematological malignancies, justifying an allo-HSCT from an alternative donor when a MRD has not been identified. It will extend the investigation of these two modalities of allo-HSCT to younger patients which are eligible to RIC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancy
* Age<55 years
* HCT-CI score ≥ 3 or non-eligible for myeloablative regimen
* Patients without a matched related donor
* Patients eligible for an allogeneic HSCT from an alternative donor
* Able to comply with the protocol
* Written informed consent
* Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen

Exclusion Criteria:

* Clinical or biological contraindication to allogeneic HSCT
* Pregnant or breast-feeding women.
* Patient considered socially or psychologically unable to comply with the treatment and the required medical follow-up.
* Severe concomitant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  the time from randomization to the time of a first occurrence of an event with death, relapse or occurrence of severe cGVHD as event and considered as censored at the time of last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Samia Harbi, MD, Principal Investigator — Institut Paoli-Calmettes; Didier Blaise, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No